CLINICAL TRIAL: NCT04724278
Title: Measuring Omalizumab Responses Using Real-world Evidence (MORRE) Study
Acronym: MORRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3475
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Asthma
Keywords: Asthma; Asthma control; Biologic; Uncontrolled Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Develop new real-world evidence indicators of worsening and improving asthma. Scientists will measure (1) steps per day, (2) duration and intensity of exercise per day, (3) sleep duration and the number of awakenings per night using Fitbit activity trackers. Scientists will measure asthma symptoms using a once-monthly custom survey delivered to participant smartphones via Twilio. Scientists may measure rescue medication use and adherence to maintenance medications using digital inhaler devices. Scientists will correlate the above measures to participant-reported significant asthma exacerbations (SAEs), lung function (FEV1), and standardized surveys (i.e. the asthma control test (ACT) and global evaluation of treatment effectiveness (GETE)(4)) collected in clinic every 3 months. Coordinators will record any medication changes or reported medication side effects.

Determine response to omalizumab therapy. After participants are placed on omalizumab therapy as part of standard medical care, scientists will determine whether and how real-world evidence can be used to gauge responses to omalizumab. Then, scientists will determine which features, or combination of features, are the best indicators of disease control in the real world.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of uncontrolled or difficult-to-treat asthma, defined as 1 course of systemic corticosteroids (e.g. oral prednisone) in the last 12 months OR an asthma control test (ACT) score less than or equal to 19 despite regular use of inhaled corticosteroids (ICS) therapy (at least 176 mcg of fluticasone/day or the equivalent) for at least 1 month prior to enrollment.
* Participants will need access to a smartphone.

Exclusion Criteria:

* Active smoking and any significant comorbid conditions that could inadvertently interfere with study results as determined by the study investigators (i.e. any terminal illness, cancer, HIV, end-stage renal disease, congestive heart failure, severe autoimmune disease or inflammatory bowel disease)
* Conditions that require bursts of oral corticosteroids
* Other significant lung diseases (cystic fibrosis, pulmonary hypertension, interstitial lung disease, pulmonary fibrosis among others)
* Other disease that may mimic asthma, including vocal cord dysfunction, hypersensitivity pneumonitis, or tracheobronchomalacia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants 18-85 years of age with moderate-to-severe asthma at the time of enrollment and eligible for omalizumab therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Asthma Control Test | Baseline and Week 52
  Standardized asthma symptom survey

SECONDARY OUTCOMES:
Change From Baseline in Significant asthma exacerbations (SAEs) | Baseline and Week 52
  A protocol-defined asthma exacerbation was defined as worsening of asthma symptoms requiring treatment with systemic corticosteroids for 3 or more days; for participants receiving long-term oral corticosteroids, an exacerbation was a 20 mg or more increase in average daily dose of oral prednisone (or a similar dose of another systemic corticosteroid). The rate of protocol-defined asthma exacerbations, normalized by subject-time at risk and computed over the 24 observation or 52-week treatment period in each treatment group.
Change From Baseline in Lung Function | Baseline and Week 52
  FEV1 % predicted pre- and post-bronchodilator FEV1 absolute (L) pre- and post-bronchodilator FVC % predicted pre- and post-bronchodilator FVC absolute (L) pre- and post-bronchodilator Bronchodilator response: % change in FEV1 after bronchodilator FEV1/FVC ratio: absolute and % predicted Aggregated measure: significant vs non significant bronchodilator reversibility. Significant reversibility defined as greater than or equal to 12% and 200mL increase in FEV1 or FVC
Global evaluation of treatment effectiveness (GETE) | Baseline and Week 52
  Standard asthma survey that is scored to assess omalizumab responders
Change From Baseline in Number of Puffs per Day of Beta Agonist Rescue Medication | Baseline and Week 52
  Number of inhalations per day averaged out over study duration Number of inhalations per night per month averaged out over study duration
Change From Baseline in Adherence of Inhaled Corticosteroids | Baseline and Week 52
  Doses taken/doses prescribed average out over study duration
Change From Baseline in Steps Per Day | Baseline and Week 52
  Steps per day average out over study duration
Change From Baseline in Duration of Exercise Per Day | Baseline and Week 52
  Minutes exercise per day average out over study duration
Change From Baseline in Intensity of Exercise Per Day | Baseline and Week 52
  Minutes exercise/day x average heart rate during the exercise
Change From Baseline in Duration of Interrupted Sleep per Night | Baseline and Week 52
  Hours of uninterrupted sleep as recorded by Fitbit device
Change From Baseline in Number of Awakenings per Night | Baseline and Week 52
  Number of awakenings per night and/or early morning awakenings as a composite score, as recorded by Fitbit
Change From Baseline in the Monthly Symptom Questionnaire Scores | Baseline and Week 52
  Each answer will be scored 1-10 points, depending on the answer, and added to create a survey score. Higher scores indicate poorer asthma control.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States